CLINICAL TRIAL: NCT05337007
Title: Impact of Protein Content of Ultraprocessed Foods on the Regulation of Energy Balance (ad Libitum Energy Intake and Energy Expenditure)
Brief Title: Impact of Protein Content of Ultraprocessed Foods on the Regulation of Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Prof. Dr. Dr. Anja Bosy-Westphal, University of Kiel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ABW-2022-HP
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: high protein foods; ultraprocessed foods; ad libitum energy intake; metabolic chamber; energy balance; macronutrient oxidation; appetite control
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: all subjects are undergoing each intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary intervention, high protein diet (Experimental): commercially available high protein ultraprocessed food items (30% protein content), cross-over design, all subjects receive all interventions
  Interventions: Other: high protein diet
- dietary intervention, moderate protein diet (Active Comparator): commercially available moderate protein ultraprocessed food items (13% protein content), cross-over design, all subjects receive all interventions
  Interventions: Other: moderate protein diet

INTERVENTIONS:
Other: high protein diet — 48 hours intervention with a 'high protein' ad libitum diet (30 % protein; 80 % commercially available ultraprocessed foods) to measure energy balance in a metabolic chamber at physical activity level of 1.45
  Arms: dietary intervention, high protein diet
Other: moderate protein diet — 48 hours intervention with a 'moderate protein' ad libitum diet (13 % protein; 80 % commercially available ultraprocessed foods) to measure energy balance in a metabolic chamber at physical activity level of 1.45
  Arms: dietary intervention, moderate protein diet

SUMMARY:
Aim of the study is to investigate the effects of high-protein, ultraprocessed foods on the regulation of energy balance in a metabolic chamber. The primary outcome parameter of the study is the energy balance (ad libitum energy intake and energy expenditure).

DETAILED DESCRIPTION:
Each of the two study weeks starts with a 3-day run-in period with controlled diet at home, following 48 hours in a metabolic chamber. On the day the participants leave the metabolic chamber, they keep a food record over the rest of the day at home.

1. week: meals containing 30 % protein (80 % ultraprocessed high-protein foods), physical activity level (PAL) 1.45, 2 intervention days in the metabolic chamber: ad libitum energy intake
2. week: meals containing 13 % protein (80 % ultraprocessed foods with moderate protein content), physical activity level (PAL) 1.45, 2 intervention days in the metabolic chamber: ad libitum energy intake

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI 19-29 kg/m2
* low-medium habitual physical activity
* women with regular menstrual cycle (during intervention in follicular phase)

Exclusion Criteria:

* smoking
* chronic illnesses (e.g. renal dysfunction)
* regular intake of medication
* food allergies / intolerances
* vegans and vegetarians
* regular high physical activity (exercise >1 hour/d)
* current weight loss diet / weight loss of >5 kg in the last 3 months
* pregnant / lactating women
* persons incapable of giving informed legal consent
* restraint eaters (according to the German version of the 'Three-Factor-Eating-Questionnaire', Stunkard und Messick (1985))

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
ad libitum energy intake | 24 hours
  ad libitum energy intake (kcal/day) of the foods consumed (breakfast, lunch, dinner, snacks)
energy expenditure | 24 hours
  measured with indirect calorimetry in a metabolic chamber (kcal/day)

SECONDARY OUTCOMES:
macronutrient oxidation | 24 hours
  measured with indirect calorimetry in a metabolic chamber (respiratory quotient, RQ)
glycemia - glucose AUC | 24 hours
  glucose AUC from continuous glucose monitoring data (mg/dL x 24 hours)
eating rate | 3 x 30 per 24 hours (during main meals)
  time to finish the meals (breakfast, lunch, dinner), (kcal/min; g/min)
oral processing behaviour (chewing) | 3 x 30 per 24 hours (during main meals)
  chews per bite, bite size, oral exposure per bite
gastric emptying | 5 hours after breakfast on first day of each intervention; intervals 15 min
  measured with 13C-octanoic acid breath test
appetite regulating hormone - ghrelin | 5 hours after breakfast on second day of each intervention; intervals 30 min
  Ghrelin concentration in plasma (15 hours AUC; pg/mL)
appetite regulating hormone - GLP-1 | 5 hours after breakfast on second day of each intervention; intervals 30 min
  Glucose Like Peptide-1 concentration in plasma (15 hours AUC; pg/mL)
appetite regulating hormone - PYY | 5 hours after breakfast on second day of each intervention; intervals 30 min
  Peptide YY concentration in plasma (15 hours AUC; pg/mL)
appetite control - subjective feelings of hunger | 5 hours after breakfast on first day of each intervention; intervals 30 min
  measured with visual analogue scales (5 hours AUC; mm x 5 hours). The scale consists of a 10 cm vertical line anchored with "not hungry at all" at the left side and with "extremely hungry" at the right side.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, PhD, MD, Principal Investigator — Institute of Human Nutrition, Kiel University
Locations (1):
- Institute of Human Nutrition, Kiel, Germany

REFERENCES:
- [Derived] Hagele FA, Herpich C, Koop J, Grubbel J, Dorner R, Fedde S, Gotze O, Boirie Y, Muller MJ, Norman K, Bosy-Westphal A. Short-term effects of high-protein, lower-carbohydrate ultra-processed foods on human energy balance. Nat Metab. 2025 Apr;7(4):704-713. doi: 10.1038/s42255-025-01247-4. Epub 2025 Mar 13. PMID 40082711